CLINICAL TRIAL: NCT06154798
Title: Effectiveness of World Digital Detox Program on Psychological Distress, Psychosocial Factors, Menopause Symptoms, and Physical Health Outcome in Women: Pragmatic Randomized Controlled Trial
Brief Title: World Digital Detox Program for Enhancing Women's Health & Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innowage Limited (Industry)
Collaborators: Zep Foundation (Unknown); Aarogyam UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Zep-WDDD-I 02
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Menopause; Menopause Related Conditions; Psychological Stress
Keywords: World Digital Detox Day Program
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- World Digital Detox Women's Health Program (Active Comparator): The intervention is a 6-week World Digital Detox Program designed to help participants reduce their dependence on digital devices and foster a healthier balance between technology use and overall well-being.
  Interventions: Behavioral: World Digital Detox Women's Health Program
- Control Group (No Intervention): Participants assigned to the control group will continue with their regular, unrestricted digital device usage throughout the 6-week study period.

INTERVENTIONS:
Behavioral: World Digital Detox Women's Health Program — World Digital Detox Women's Health Program incorporates gradual steps, including mindfulness exercises, setting boundaries on digital usage, decluttering digital spaces, promoting offline connections, and encouraging mindful technology use.
  Arms: World Digital Detox Women's Health Program

SUMMARY:
The concept of a digital detox, involving a deliberate reduction or elimination of digital device usage, has emerged as a potential strategy to mitigate the adverse effects of technology on mental and physical well-being. However, the specific effects of a structured digital detox program on psychological distress, psychosocial factors, menopause symptoms, and overall physical health in a community context remain underexplored.

This study seeks to address this gap by conducting a real-world trial, examining the impact of a digital detox program tailored for women. By delving into the intricacies of how digital technology interacts with the unique challenges faced by women, this research aims to contribute valuable insights into the development of real-world-driven interventions that promote the holistic well-being of women in the digital age.

DETAILED DESCRIPTION:
Excessive screen time and social media use during menopause pose multifaceted challenges. Prolonged exposure to screens can disrupt sleep patterns and exacerbate existing sleep disturbances, impacting the hormonal balance crucial for menopausal women. Social media's potential to induce stress, anxiety, and negative self-perception adds an emotional layer, while sedentary screen-related behavior may contribute to physical health concerns such as weight gain and decreased bone density, issues already pertinent to menopausal women. The impact on interpersonal relationships, cognitive function, body image, and time management further complicates the landscape, highlighting the need for mindful strategies to navigate the intersection of menopause and digital habits.

The World Digital Detox Program, developed by the Zep Foundation, takes a comprehensive approach to address challenges associated with increased screen and social media use, extending its focus to encompass the unique challenges faced by women during menopause. The concept of a digital detox, involving a deliberate reduction or elimination of digital device usage, has emerged as a potential strategy to mitigate the adverse effects of technology on mental and physical well-being.

The overarching aim is to enhance the comprehensive well-being of women in the digital era, going beyond addressing broad concerns of prolonged screen usage. The focus is on tailoring interventions to meet the distinct needs of women navigating the complexities of menopause. This involves incorporating practices such as breathwork, exercise, dietary adjustments, and overall well-being strategies, ensuring a holistic approach that considers the unique challenges and requirements of women during this life stage.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal staging: perimenopause or postmenopausal as per STRAW definitions
* Speak, read, and write in English sufficiently to comprehend materials in group treatment.

Exclusion Criteria:

* Participants who are severely depressed
* Need for acute treatment
* Participants with Psychotic Disorders, or current Substance Dependence.
* On Hormonal Replacement Therapy or intent to in next 3-months

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women in Menopause stage
Enrollment: 73 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Menopausal Health-Related Quality of Life | Baseline to 6-weeks post intervention
  Menopausal Health-Related Quality of Life -38 items questionnaire score on a 4-point or binary scale covering 4 major domains (physical health, mental health, life satisfaction, and social involvement) of a woman's health during the menopausal transition

SECONDARY OUTCOMES:
Clinical Global Impression Scale (CGI) | Baseline to 6-weeks post intervention
  The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients).
Client Satisfaction Questionnaire (CSQ) | Baseline to 6-weeks post intervention
  CSQ-8 items scores on a 4-point scale (possible range from eight to 32, where a higher score indicates a higher level of overall satisfaction with services,

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Chaudhari, PhD, Study Director — World Digital Detox Day, Zep Foundation; Neha Sharma, PhD, Study Chair — Aarogyam UK
Locations (1):
- World Digital Detox Day, Mumbai, Maharashtra, India